CLINICAL TRIAL: NCT00986973
Title: A Pilot Study of FDG PET Findings in Patients With Phenylketonuria Before and After BH4 Supplementation
Brief Title: Fluorodeoxyglucose Positron Emission Tomography (FDG PET) Findings in Patients With Phenylketonuria Before and After KUVAN Therapy
Acronym: PKU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 09-007154
Record Dates: First submitted 2009-09-28; First posted 2009-09-30 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Phenylketonuria
Keywords: PKU; BH4; KUVAN; PET scan; Neurodevelopment
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sapropterin (KUVAN) (Experimental): All subjects will receive Sapropterin (KUVAN) therapy at a dose of 20/mk/kg/day for four months.
  Interventions: Drug: Sapropterin

INTERVENTIONS:
Drug: Sapropterin — All subjects will receive 20 mg/kg/day Sapropterin (KUVAN) for four months. Subjects will be examined with fluorodeoxyglucose positron emission tomography (FDG-PET) brain imaging, physical and neurological exam, blood tests for phenylalanine (Phe) and tyrosine levels, and neuropsychological testing before and 4 months after KUVAN therapy. Subjects Phe and tyrosine levels will be monitored weekly during the study and subjects will keep 3-day diet records to allow for calculation of Phe intake.
  Other Names: KUVAN; BH4

SUMMARY:
The aim of this pilot study is to determine if there are any changes in brain glucose metabolism in the gray matter of patients with Phenylketonuria (PKU) and whether administration of Sapropterin (KUVAN) therapy can improve such deficits.

DETAILED DESCRIPTION:
Phenylketonuria (PKU) is an autosomal recessive disorder resulting from a deficiency of phenylalanine hydroxylase, which converts phenylalanine to tyrosine. Phenylalanine hydroxylase is one of the three aromatic amino acid hydroxylases that utilizes tetrahydrobiopterin (BH4) as cofactor. The published reports indicate that there is altered energy metabolism in the brain of patients with PKU. Phenylalanine and its metabolites appear to impair several aspects of brain energetics including: (1) Inhibition of glucose uptake; (2) diminished glycosylation of cytoskeletal proteins; (3) Inhibition of pyruvate kinase; and (4) reduced flux through the glycolysis. Studies in vivo with magnetic resonance spectroscopy have demonstrated phenylalanine-responsive abnormalities in cerebral energy metabolism.

Positron Emission Tomography (PET) scanning with fluorodeoxyglucose (FDG-PET) is a non-invasive method that measures regional glucose metabolic rate with high resolution and absolute quantitation. To date this technology has been used only for single case reports or the investigation of white matter abnormalities in small numbers of patients with PKU.

The aim of this pilot study is to determine if there are any changes in brain glucose metabolism in the gray matter of patients with PKU and whether Sapropterin (KUVAN) can improve such deficits. This study will also elucidate the relationship between hyperphenylalaninemia, phenylalanine intake in diet, altered brain glucose handling and the neurocognitive profile of the patients with PKU before and after KUVAN therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females over the age of 18 years
2. Subject must be able to give independent informed consent
3. Girls must have a negative urine pregnancy test and must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or an oral contraceptive, for the duration of the study.
4. Subject must have a confirmed diagnosis of PKU
5. Subjects with Phenylalanine (Phe) levels over 10 mg/dL
6. Subjects naïve to KUVAN therapy or has not received KUVAN in the 6 months before screening

Exclusion Criteria:

1. Pregnancy
2. Cognitive deficits resulting from physical trauma (e.g. subject with history of severe birth trauma).
3. Neurologic comorbidities including a history of a stroke or a seizure disorder.
4. Laboratory abnormalities that indicate clinically significant hepatic disease Aspartate aminotransferase (AST)> 2.0 times the upper limit of normal, Alanine transaminase (ALT) > 2.0 times the upper limit of normal, Prothrombin Time (PT) > 2.0 times the upper limit of normal, Partial Thromboplastin Time(PTT) > 2.0 times the upper limit of normal
5. Subjects using medications such as steroids, insulin and glucagons that may interfere with the results of PET scan.
6. Subjects using medications that inhibit folate metabolism such as methotrexate
7. Subjects using medications known to affect nitric oxide-mediated vasorelaxation.
8. Subjects using Levodopa
9. Treatment with KUVAN in the past 6 months before study entry.
10. Treatment with any investigational product in the last 90 days before study entry

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Can Ficicioglu, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia,University of Pennsylvania
Locations (1):
- Children's Hospital of Philadelphia, Section of Metabolism,PKU program, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Classical PKU who were being followed at Children's Hospital of Philadelphia were recruited between 2010 and 2011. Study participation was presented during routine clinic visits and interested subjects were screened for eligibility. A flier was posted on PKU support group websites help recruit additional subjects.
Pre-assignment Details: Six adults (4 male and 2 females) were interested in participating in the study, each signed informed consent forms and were screened for eligibility. All six were enrolled.
Groups:
- Sapropterin (KUVAN): All subjects received 20 mg/kg/day Sapropterin (KUVAN) for four months. Subjects were examined with fluorodeoxyglucose positron emission tomography (FDG-PET) brain imaging, physical and neurological exam, blood tests for phenylalanine (Phe) and tyrosine levels, and neuropsychological testing before and 4 months after KUVAN therapy. Subjects' Phe and tyrosine levels were monitored weekly during the study and subjects kept 3-day diet records to allow for calculation of Phe intake.
Period: Overall Study
Arm/Group | Sapropterin (KUVAN)
Started | 6
Completed | 5 (One subject was withdrawn from the study due to poor compliance with KUVAN therapy.)
Not Completed | 1
Not completed — Withdrawn by study team | 1

BASELINE CHARACTERISTICS:
Groups:
- Sapropterin (KUVAN): All subjects received 20 mg/kg/day KUVAN for four months.
Arm/Group | Sapropterin (KUVAN)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Plasma Phenylalanine Level (mg/dl)
Description: Plasma phenylalanine level (mg/dl) served as the primary means of evaluating brain glucose metabolism before and after sapropterin (KUVAN) therapy. Blood tests for phenylalanine levels (Phe) were collected before and 4 months after sapropterin (KUVAN) therapy. All subjects received KUVAN at a dose of 20/mg/kg/day for four months. The goal was to estimate the change in blood glucose metabolism after treatment with Sapropterin (if any), with the hypothesis that treatment would decrease plasma Phe levels.
Time Frame: Measurements were obtained at the beginning and conclusion of each study period (baseline and 4 months)
Population: 1 subject was withdrawn from the study due to poor compliance with KUVAN therapy.
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Sapropterin (KUVAN) Therapy: All subjects received KUVAN at a dose of 20/mg/kg/day for four months. Blood Phe levels were measured drawn before therapy and 4 months after starting therapy.
Arm/Group | Sapropterin (KUVAN) Therapy
Number analyzed (Participants) | 5
mg/dl
  Phe Level Before KUVAN Therapy (mg/dl) | 18.0 (18.95)
  Phe Level 4 Months After KUVAN Therapy (mg/dl) | 17.2 (16.35)
Statistical Analysis 1: Comparison: Sapropterin (KUVAN) Therapy; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

2. Secondary Outcome: Hopkins Verbal Learning Test (HVLT) Total Recall
Description: The Hopkins Verbal Learning Test-Revised (HVLT) is a neuropsychological test designed to assess verbal memory. The test consists of 12 nouns (targets) with four words drawn from each of three semantic categories. Raw scores are derived for Total Recall (across three learning trials), Delayed Recall (after 20-25 minute delay), Retention (% retained), and a Recognition Discrimination Index (true positives minus false positives). The maximum total for each recall trial (Learning Trials 1 to 3, Delayed Recall Trial 4) is 12. Raw scores are converted to "T-scores" by means of age-based tables provided in test manual (T-scores can go from 0 - 100, with higher scores correlating with higher verbal memory function). Median HVLT Total Recall and HVLT Delayed Recall T-scores at baseline and 4 months after Sapropterin therapy were compared.
Time Frame: Measures were obtained at the beginning and conclusion of each study period (baseline and 4 months)
Population: 1 Subject was withdrawn from the study due to poor compliance with KUVAN therapy and did not complete all HVLT assessments.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Sapropterin (KUVAN)
Number analyzed (Participants) | 5
units on a scale
  HVLT Total Recall T-Score at Baseline | 51 [27.5 to 57]
  HVLT Total Recall T-Score Post-Sapropterin | 53 [29 to 54]
Statistical Analysis 1: Comparison: Sapropterin (KUVAN); Test type: Superiority or Other; p = 0.82, Friedman test; Non-parametric test was used to examine neuropsychological outcomes

3. Secondary Outcome: Hopkins Verbal Learning Test (HVLT) Delayed Recall
Description: as for outcome 2
Time Frame: Measures were obtained at the beginning and conclusion of each study period (baseline and 4 months)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Sapropterin (KUVAN)
Number analyzed (Participants) | 5
units on a scale
  HVLT Delayed Recall T-Score at Baseline | 47 [25 to 75]
  HVLT Delayed Recall T-Score Post-Sapropterin | 49 [33.50 to 56.5]
Statistical Analysis 1: Comparison: Sapropterin (KUVAN); Test type: Superiority or Other; p = 0.46, Friedman test; Non-parametric test was used to examine neuropsychological outcomes

4. Secondary Outcome: Paced Auditory Serial Addition Task (PASAT)
Description: The Adapted Paced Auditory Serial Addition Task (PASAT) is a measure of cognitive function that specifically assesses auditory information processing speed and flexibility, as well as calculation ability. For Rates #1 and #2, single digits are presented every 3 seconds and the patient must add each new digit to the one immediately prior to it. The score for PASAT is the total number of correct answers (out of 60, for a total possible score ranging from 0-60 with higher score preferred as it indicates higher auditory processing speed) for each trial. All scores are expressed as "z-scores" which are generated based on norms for 101 healthy adults, with separate norms for <12 years of education versus >12years of education. Using a reference population as a basis of comparison, the "z-score" is the number of standard deviations the score is above (positive) or below (negative) the mean of the reference population (zero). Possible z-scores lie on a continuous scale.
Time Frame: Measures were obtained at the beginning and conclusion of each study period (baseline and 4 months)
Population: 1 Subject was withdrawn from the study due to poor compliance with KUVAN therapy and did not complete all PASATassessments.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Sapropterin (KUVAN)
Number analyzed (Participants) | 5
units on a scale
  PASAT Z-score at Baseline | 0.4700 [-0.6375 to 0.7450]
  PASAT Rate #1 Z-score Post-Sapropterin | 0.94 [0.8075 to 1.1775]
Statistical Analysis 1: Comparison: Sapropterin (KUVAN); Test type: Superiority or Other; p = 0.071, Friedman test; Non-parametric test was used to examine neuropsychological outcomes

5. Secondary Outcome: Symbol-Digit Modalities Test (SMTD)
Description: The symbol-digit modalities test (SDMT) was developed to identify individuals with neurological impairment. The SDMT requires individuals to identify nine different symbols corresponding to the numbers 1 through 9, and to practice writing the correct number under the corresponding symbol. Then they manually fill the blank space under each symbol with the corresponding number. A second oral administration is then completed. The participant is given a blank copy of the test and asked to state the correct number for each corresponding symbol. The participant is given 90 s to complete each of these administrations. A written and oral score is calculated by totaling the number of correct answers for each section. The score is the number of correctly coded items from 0-110 in 90 seconds, with a higher score representing less neurological impairment with respect to attention, scanning abilities and motor skills. The total raw score was used for purposes of this study.
Time Frame: Measures were obtained at the beginning and conclusion of each study period (baseline and 4 months)
Population: 1 Subject was withdrawn from the study due to poor compliance with KUVAN therapy and did not complete all SMTD assessments.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Sapropterin (KUVAN)
Number analyzed (Participants) | 5
units on a scale
  SDMT Raw Score at Baseline | 63 [38 to 75.50]
  SDMT Raw Score Post-Sapropterin | 79 [41.50 to 80.50]
Statistical Analysis 1: Comparison: Sapropterin (KUVAN); Test type: Superiority or Other; p = 0.25, Friedman test; Non-parametric test was used to examine neuropsychological outcomes

6. Secondary Outcome: Wechsler Adult Intelligence Scale (WAIS-IV)-Digit Span
Description: The Wechsler Adult Intelligence Scale (WAIS) is a test designed to measure intelligence in adults and older adolescents. It is composed of 10 core subtests and five supplemental subtests, with the 10 core subtests comprising the Full Scale intelligence quotient (IQ). Contained within the WAIS is an assessment of digit-coding which consists of nine digit-symbol pairs followed by a list of digits. Under each digit the subject should write down the corresponding symbol as fast as possible. The number of correct symbols within the allowed time (e.g. 90 or 120 sec) is measured, with a higher score representative of a higher performance component of IQ/intelligence.
Time Frame: Measures were obtained at the beginning and conclusion of each study period (baseline and 4 months)
Population: 1 Subject was withdrawn from the study due to poor compliance with KUVAN therapy and did not complete all WAIS-IV assessments.
Measure: Median (Inter-Quartile Range); unit: Number of correct symbols
Arm/Group | Sapropterin (KUVAN)
Number analyzed (Participants) | 5
Number of correct symbols
  WAIS-IV Digit Span Raw Score at Baseline | 33 [19.50 to 35.50]
  WAIS-IV Digit Span Raw Score after Sapropterin | 37 [19.50 to 38.0]
Statistical Analysis 1: Comparison: Sapropterin (KUVAN); Test type: Superiority or Other; p = 0.050, Friedman test; Non-parametric test was used to examine neuropsychological outcomes

7. Secondary Outcome: Delis-Kaplan Executive Function System Verbal Fluency Subtest (D-KEFS)
Description: The Delis-Kaplan Executive Function System (D-KEFS) is a neuropsychological test is used to measure a variety of verbal and nonverbal executive functions for both children and adults. Among the 9 subtests is the Verbal Fluency Test which measures letter fluency, category fluency, and category switching. Verbal Fluency Test. This subtest requires an individual to randomly generate words based upon given parameters (ex., as words beginning with the letter F) and the believed areas of executive function assessed are cognitive flexibility, response inhibition, and verbal fluency. Raw scores are calculated based on the number of correct answers, which are then converted to scaled scores with a mean of 10 and standard deviation of 3. Higher scaled score represents a higher level of executive verbal and nonverbal function.
Time Frame: Measures were obtained at the beginning and conclusion of each study period (baseline and 4 months)
Population: 1 Subject was withdrawn from the study due to poor compliance with KUVAN therapy and did not complete all assessments.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Sapropterin (KUVAN)
Number analyzed (Participants) | 5
units on a scale
  Scaled D-KEFS Fluency Score at baseline | 10 [5 to 10]
  Scaled D-KEFS Fluency Score after Sapropterin | 11 [5 to 12.50]
Statistical Analysis 1: Comparison: Sapropterin (KUVAN); Test type: Superiority or Other; p = 0.34, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from baseline through the end of study treatment (4 months).
Groups:
- Sapropterin (KUVAN) Therapy: All subjects will received KUVAN therapy 20 mg/kg/day for four months.
Arm/Group | Sapropterin (KUVAN) Therapy
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Due to small sample size, the statistical power of this study is low. While it is useful in exploring potential trends, the results of this pilot study should be cautiously interpreted. Further studies with a larger sample of subjects are needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No